CLINICAL TRIAL: NCT00573391
Title: A Phase III Study for Patients Relapsing or Progressing After Autologous Transplantation on Total Therapy 2 (TT2, UARK 98-026): Bortezomib, Thalidomide and Dexamethasone Versus Bortezomib, Melphalan, and Dexamethasone
Brief Title: Study of Multiple Myeloma Patients Relapsing or Progressing After Autologous Transplantation on Total Therapy 2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: University of Arkansas (Other)
Responsible Party: Bart Barlogie, MD, PhD, University of Arkansas for Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-05
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Results first posted 2011-08-12 (Estimated); Last update posted 2011-08-12 (Estimated); Status verified 2011-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Thalidomide; Dexamethasone; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VTD = Velcade, Thal, and Dex (Experimental): VTD = Velcade, Thalidomide, and Dexamethasone
  Interventions: Drug: Velcade, Thalidomide, and Dexamethasone
- VMD = velcade, melphalan, and dex (Experimental): VMD = velcade, melphalan, and dexamethasone
  Interventions: Drug: Velcade, Melphalan, and Dexamethasone

INTERVENTIONS:
Drug: Velcade, Thalidomide, and Dexamethasone — Velcade - Into vein (IV) Days 1, 4, 8, 11
  Yr 1: Every 28-35 days-12 cycles
  Yr 2: Every 8-10 weeks- 6 cycles
  Thalidomide - By Mouth Days 1-28
  Yr 1: Every 28-35 days-12 cycles
  Yr 2: Every 8-10 weeks- 6 cycles
  Arms: VTD = Velcade, Thal, and Dex
Drug: Velcade, Melphalan, and Dexamethasone — Velcade - Into vein (IV) Days 1, 4, 8, 11
  Yr 1: Every 28-35 days-12 cycles
  Yr 2: Every 8-10 weeks- 6 cycles
  Arms: VMD = velcade, melphalan, and dex

SUMMARY:
This study is being done to find out if the combination of VelcadeTM with melphalan and dexamethasone (VMD) will be as effective, or even more effective as it is in combination with thalidomide and dexamethasone (VTD).

DETAILED DESCRIPTION:
A new drug (bortezomib [VelcadeTM PS-341]) has been shown in recent studies to be effective in subjects with advanced multiple myeloma. There is also research that shows this drug may be even more effective when used in combination with other drugs that have been used to treat myeloma for many years (melphalan, thalidomide, and dexamethasone). This study is being done to find out if the combination of VelcadeTM with melphalan and dexamethasone (VMD) will be as effective, or even more effective as it is in combination with thalidomide and dexamethasone (VTD).

ELIGIBILITY:
Inclusion Criteria:

* History of histologically documented MM previously enrolled on UARK 98-026 with relapsed or progressive disease after at least one autologous transplant.
* Patient has measurable disease in which to capture response, defined as:
* Serum M-protein level > 1.0 gm/dl (10.0 g/L) measured by serum protein electrophoresis or immunoglobulin electrophoresis
* Urinary M-protein excretion > 200 mg/24 hrs
* Bone marrow plasmacytosis of > 30percent by bone marrow aspirate and/or biopsy
* Serum Free Light Chains (By the Freelite test) > 10 mg/dL with an abnormal kappa/lambda ration.
* 50percent increase in size of lytic and/or focal lesions or development of new lesions recognized by radiographic studies.
* Performance status of 2 as per SWOG scale, unless PS of 3-4 based solely on bone pain.
* Patients must have a platelet count 50,000/mm3, unless the low platelet count is due to documented (>30 percent) extensive myeloma infiltration of the bone marrow.
* Patients must have adequate renal function defined as serum creatinine < 2.5 mg/dl.
* Patients must have adequate hepatic function defined as serum transaminases and direct bilirubin < 2 x the upper limit of normal.
* Pregnant or nursing women may not participate. Women of childbearing potential must have a negative pregnancy documented within one week of registration. Women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Male or female adults of at least 18 years of age.
* Patients must have signed and IRB-approved written informed consent form and demonstrate willingness to meet follow-up schedule and study procedure obligations
* > 5 x 106 CD34 cells/kg in storage strongly desired, but not mandated

Exclusion Criteria:

* Not previously enrolled on UARK 98-026.
* Has received salvage therapy after coming off UARK 98-026.
* Evidence of POEMS Syndrome..
* Significant neurotoxicity interfering with ADL.
* Platelet count < 50,000/mm3
* Clinically significant hepatic dysfunction as noted by bilirubin or AST >3 times the upper normal limit or clinically significant concurrent hepatitis.
* New York Hospital Association (NYHA) Class III or Class IV heart failure.
* Myocardial infarction within the last 6 months.
* Truly non-secretory MM (no increase in serum free-light chains) in the absence of bone marrow plasmacytosis and MRI-defined focal lesions with CT-FNA-proven MM
* Uncontrolled, active infection requiring IV antibiotics.
* Patients with a history of treatment for clinically significant ventricular cardiac arrhythmias.
* Poorly controlled hypertension, diabetes mellitus, or other serious or psychiatric illness that could potentially interfere with the completion of treatment according to this protocol.
* Pregnant or potential for pregnancy. Women of childbearing potential will have a pregnancy test at screening, and will be required to use a medically approved contraceptive method. Pregnancy testing will be performed prior to administration of each dose of study drug.
* Breast-feeding women may not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Barlogie, MD, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Usmani SZ, Sexton R, Hoering A, Heuck CJ, Nair B, Waheed S, Al Sayed Y, Chauhan N, Ahmad N, Atrash S, Petty N, van Rhee F, Crowley J, Barlogie B. Second malignancies in total therapy 2 and 3 for newly diagnosed multiple myeloma: influence of thalidomide and lenalidomide during maintenance. Blood. 2012 Aug 23;120(8):1597-600. doi: 10.1182/blood-2012-04-421883. Epub 2012 Jun 6. PMID 22674807

RESULTS

PARTICIPANT FLOW:
Groups:
- Velcade, Thalidomide, and Dexamethasone: Velcade 1.0 mg/m^2 Velcade 1.3 mg/m^2 D1,4, 8, 11 (x 6 cycles, then 1.0 mg/m^2 (for cycles 7-12) Thalidomide 100 mg D1-28 Dexamethasone 20 mg D1-4 and 8-11
- VMD With Melphalan Dose Escalation: VMD:
  Velcade 1.3 mg/m^2 D1, 4, 7, 10 (x6 mo, then 1.0 mg/m^2) Melphalan 4 (6, 8, 10) mg/m^2 D1, 4, 7, 10 dose escalation Dexamethasone 20 mg 1-4 and 7-10
Period: Overall Study
Arm/Group | Velcade, Thalidomide, and Dexamethasone | VMD With Melphalan Dose Escalation
Started | 3 | 2
Completed | 0 | 0
Not Completed | 3 | 2
Not completed — study stopped | 2 | 2
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Velcade, Thalidomide, and Dexamethasone | VMD With Melphalan Dose Escalation | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Participant Survival With Velcade/Melphalan/Dexamethasone Treatment vs. Participant Survival With Velcade/Thalidomide/Dexamethasone Treatment
Description: due to low accrual rates, no analyses was done to compare the new combination of Velcade/Melphalan/Dexamethasone vs. Velcade/Thalidomide/Dexamethasone
Time Frame: 24 months
Measure: Number; unit: Participant
Arm/Group | Velcade, Thalidomide, and Dexamethasone | VMD With Melphalan Dose Escalation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Velcade, Thalidomide, and Dexamethasone | VMD With Melphalan Dose Escalation
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/5
Other Adverse Events (participants affected / at risk) | 2/5 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velcade, Thalidomide, and Dexamethasone (N=5) | VMD With Melphalan Dose Escalation (N=5)
fever (General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velcade, Thalidomide, and Dexamethasone (N=5) | VMD With Melphalan Dose Escalation (N=5)
secondary pulmonary hypertension (Cardiac disorders) | 1 (1) | 0 (0)
pneumonia (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
early termination due to low accrual, no analyses

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes